CLINICAL TRIAL: NCT02100137
Title: Women With Asymptomatic Endometrial Hyperplasia
Acronym: FAME-ENDO
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, LHefler, Associate Professor, Medical University of Vienna
Other Study IDs: AGO 12; AGO Austria (Other: AGO Austria)
Record Dates: First submitted 2012-03-05; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with endometrial hyperplasia
  Interventions: Other: vaginal ultrasound

INTERVENTIONS:
Other: vaginal ultrasound — vaginal ultrasound performed at a routine gyn examination

SUMMARY:
The purpose of this study is to evaluate the clinical meaning of an endometrial hyperplasia diagnosed using a vaginal ultrasound during routine gynecological examination.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic women with endometrial hyperplasia diagnosed using a vaginal ultrasound

Exclusion Criteria:

* postmenopausal bleeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: asymptomatic women with endometrial hyperplasia diagnosed using a vaginal ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2006-09; Primary Completion 2010-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of invasive endometrial cancers | Participants will be followed for the duration of hospital and until the results of the final histology from the endometrial biopsy are completed, for an expected average of 10 days

SECONDARY OUTCOMES:
Number of women with atypical endometrial hyperplasia | Participants will be followed for the duration of hospital and until the results of the final histology from the endometrial biopsy are completed, for an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hefler, Associate Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria